CLINICAL TRIAL: NCT00382551
Title: The Effect of Alcohol and Polyphenolic Compounds on Endothelial Function
Brief Title: The Effect of Beer, Red Wine and Fruit Juice on Blood Vessel Function in Persons With Cardiovascular Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: VN-20060043
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Heart Disease
Keywords: Alcohol; Red wine; Endothelial function; Flow-mediated vasodilation; Cardiovascular disease
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases

INTERVENTIONS:
Behavioral: Moderate daily consumption of Red wine
Behavioral: Moderate daily consumption of beer
Behavioral: Moderate consumption of fruit juice rich in polyphenolics

SUMMARY:
To study the effect of red wine, beer and fruit juice on endothelial function in patients with coronary Heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Men or postmenopausal women with stable coronary heart disease
* Coronary heart disease should be verified by coronary angiography with at least 50% stenosis in at least one coronary vessel.

Exclusion Criteria:

* Patients with myocardial infarction within the last tree months
* Persons with a present or earlier alcohol abuse
* Persons with a present or earlier drug abuse
* Person with malign disease
* Persons, that we consider unsuitable to carry through the examines.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Changes in flow-mediated vasodilation after 2 weeks intervention compared with baseline

SECONDARY OUTCOMES:
Lipid status after 2 weeks intervention compared with baseline
Effects in Coagulation factors after 2 weeks intervention
Effects on markers of inflammation after 2 weeks intervention
Effects on markers of endothelial function after 2 weeks intervention
Changes in the overall antioxidant activity in plasma after 2 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Erik B Schmidt, Professor, Study Director — Department of Cardiology, Aalborg Hospital , Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aalborg Hospital, Science and Innovation Center, Aalborg, Aalborg, Denmark